CLINICAL TRIAL: NCT06803394
Title: Hearing Health Equity Through Accessible Research and Solutions for Korean Americans
Acronym: K-HEARS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00406742; R01DC019686 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Age-related Hearing Impairment; Personal Communication; Hearing Impairment; Hearing Loss; Community-dwelling Seniors; Korean
MeSH Terms: conditions — Communication; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Site (Experimental): Study site assigned to immediate treatment of K-HEARS intervention
  Interventions: Behavioral: K-HEARS Intervention; Device: K-HEARS Sound Amplifier Intervention
- Delayed Treatment Site (Placebo Comparator): Study site assigned to 6-month delayed treatment of K-HEARS intervention
  Interventions: Behavioral: K-HEARS Intervention; Device: K-HEARS Sound Amplifier Intervention

INTERVENTIONS:
Behavioral: K-HEARS Intervention — Tailored aural rehabilitation for participant and care partner
Device: K-HEARS Sound Amplifier Intervention — Tailored fitting and programming of a personal sound amplifier. This will be accompanied by a component of aural rehabilitation.

SUMMARY:
The objective of this study is to test the effect of a community-delivered, affordable, and accessible hearing care intervention on improving communication function and health-related quality of life among older Korean Americans (KA) and the older Korean American's care partners that integrates a low-cost over-the-counter amplification device and hearing rehabilitation in comparison to a 6-month delayed treatment group through a cluster randomized controlled study.

ELIGIBILITY:
PARTICIPANT CRITERIA Participant inclusion criteria

* Self-identified as first-generation KA in the target region
* Age 60 years or older
* Has a communication partner who lives in the same household or has at least weekly interactions
* Screening audiometry Pure-tone audiometry (PTA)1,2,4 kilohertz (kHz) >25 decibel (dB) hearing loss (HL) in better ear
* Hearing handicap as measured by HHIE-S score >=8 Participant exclusion criteria
* Current use of hearing aid
* Medical contraindications to use amplification device (e.g., draining ear)
* Plan to move from the area within 6 months
* Active treatment for a terminal illness or in hospice

COMMUNICATION PARTNER CRITERIA Communication Partner inclusion criteria

* Age 18 years or older
* Able to read and speak Korean
* Lives with the older adult or has at least weekly interactions Communication Partner exclusion criteria
* Plan to move from the area within 6 months
* Active treatment for a terminal illness or in hospice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-02-09 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Hearing Handicap Inventory for the Elderly (HHIE-S) score | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  Score range 0-40. 0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap.

SECONDARY OUTCOMES:
Third Party Disability as assessed by the Significant Other Scale for Hearing Disability (SOS-HEAR) | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  Third-party disability will be measured in communication partners using the Significant Other Scale for Hearing Disability (SOS-HEAR). Score range 0-104, with higher score more disability.
Relationship Quality as assessed by the Mutuality Scale | Baseline, 6 months post-intervention (Immediate Group). 6 months post-baseline (Delayed Group)
  Relationship quality will be measured using the Mutuality Scale among participants and communication partners. Score range 0-60, with higher score better relationship quality.

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD,RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States